CLINICAL TRIAL: NCT00798980
Title: Scandinavian Mirena Insertion Nulliparous Trial of an Observational Study.
Brief Title: Scandinavian Mirena Insertion Nulliparous Trial.
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Schering Pharma AG
Other Study IDs: 14015; MA0710SE; SCAN 68/06; 2006/0601120
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Nulliparous
Keywords: Mirena; Nulliparous; Intrauterine Devices
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1
  Interventions: Drug: Mirena (BAY86-5028)

INTERVENTIONS:
Drug: Mirena (BAY86-5028) — Nulliparous Women

SUMMARY:
In this non-interventional study we investigate the nulliparous women individual evaluation of the insertion procedure of LNG-IUD and the follow-up period of 3 months post insertion.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women Mirena insertion planned as contraceptive method

Exclusion Criteria:

* Ongoing or suspected pregnancy;
* Ongoing or recidivating genital infection;
* Cervicitis;
* Cervical dysplasia;
* Malignancy in uterus or cervix;
* Confirmed or suspected hormone sensitive neoplasia including breast cancer
* Undiagnosed abnormal uterine bleeding;
* Uterine anomaly including myoma if the cavity of the uterus is restricted;
* Conditions that cause increased risk of infections;
* Acute liver disease or liver tumour;
* Allergy to the active substance or any component of the IUD

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic Patients
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the insertion procedure of Mirena in nulliparous women | At the insertion time point

SECONDARY OUTCOMES:
Pain | At the insertion time point
Continuation rate | 12-16 weeks post insertion
Bleeding Pattern | 12-16 weeks post insertion
Satisfaction | 12-16 weeks post insertion

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Sweden

REFERENCES:
- [Result] Marions L, Lovkvist L, Taube A, Johansson M, Dalvik H, Overlie I. Use of the levonorgestrel releasing-intrauterine system in nulliparous women--a non-interventional study in Sweden. Eur J Contracept Reprod Health Care. 2011 Apr;16(2):126-34. doi: 10.3109/13625187.2011.558222. PMID 21417562